CLINICAL TRIAL: NCT04253860
Title: Effect of Transcutaneous Electrical Nerve Stimulation on Pain percepción and Serum Inflammatory Markers in Patients With Peripheral Diabetic Neuropathy
Brief Title: Effect of Transcutaneous Electrical Nerve Stimulation in Diabetic Neuropathy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to pandemic od COVID-19, was difficult recruit patients
Sponsor: Centro Universitario de Tonalá (Other)
Collaborators: University of Guadalajara (Other); Diabetes sin Complicaciones S.A de C.V, Mexico (Unknown)
Responsible Party: Principal Investigator, Arieh Roldán Mercado Sesma, Investigator, Centro Universitario de Tonalá
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TENS-ND-2018
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Diabetic Neuropathy Peripheral
Keywords: Diabetic neuropathy peripheral; diabetic complications; TENS; Neuropathic treatments
MeSH Terms: conditions — Diabetes Complications

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, clinical trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS (Experimental): Transcutaneous electrical neurostimulation will be applied for 30 minutes three times a week during 90 days
  Interventions: Device: Transcutaneous electrical neurostimulation
- Sham (Sham Comparator): A sham comparator will be applied for 30 minutes three times a week during 90 days. The device does not emit electrical impulses
  Interventions: Device: Transcutaneous electrical neurostimulation

INTERVENTIONS:
Device: Transcutaneous electrical neurostimulation — Sessions of 30 minutes of TENS will be applied three times a week during 90 days

SUMMARY:
Double-blind, randomized, placebo-controlled, clinical trial. Patients with diabetic neuropathy will be randomly assigned to treatment with either TENS or TENS sham three times a week during 90 days. Clinical determinations are: pain, levesls of TNF-alpha, IL-6 and RPC-us

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic of type 2 diabetes > 10 years
* Diagnostic of peripheral diabetic neuropathy less than 5 years
* HbA1C > 6.5 and < 9%
* Plasmatic glucose >140 mg/dL and lees than 350 mg/dL
* Informed consent signed

Exclusion Criteria:

* Use of implanted pacemaker or heart defibrillator
* Implanted brain stimulator
* History of alcohol abuse
* Use of NSAID, stereoids
* Subjects with wounds, ulcers in legs
* Subjects with hepatic, renal o neurologic diseases

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Pain perception | Change from Baseline Pain perception at 90 days
  Evaluation of neuropathic pain evaluated with VAS

SECONDARY OUTCOMES:
Tumoral Necrosis Factor Alpha | Change from Baseline serum levels of TNF-alpha at 90 days
  Serum levels of TNF-alpha
Interleukin-6 | Change from Baseline serum levels of IL-6 at 90 days
  Serum levels of IL-6
C Reactive Protein ultra-sensible | Change from Baseline serum levels of CRP-us at 90 days
  Serum levels of CRP-us

CONTACTS AND LOCATIONS:
Overall Officials: Arieh R Mercado Sesma, PhD, Principal Investigator — Salud Enfermedad como proceso individual, CUTonalá, Universidad de Guadalajara
Locations (1):
- University of Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No